CLINICAL TRIAL: NCT06614361
Title: Community-based Behavioral Intervention to Increase COVID-19 and Influenza Vaccination for African American/ Black and Latino Persons: An Optimization Randomized Controlled Trial
Brief Title: Community-based Behavioral Intervention to Increase Vaccination Using MOST
Acronym: NCAP2
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: terminated by NIH
Sponsor: New York University (Other)
Collaborators: Northern Manhattan Improvement Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: IRB-FY2025-9851
Record Dates: First submitted 2024-09-25; First posted 2024-09-26 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-03

CONDITIONS: COVID 19; Influenza
Keywords: COVID-19; influenza; vaccination
MeSH Terms: conditions — COVID-19; Influenza, Human | interventions — Influenza Vaccines; Vaccination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Experimental Condition 1 (Experimental): Core session
  Interventions: Behavioral: Health education on COVID and flu vaccination
- Experimental Condition 12 (Experimental): Core session, nurse-led SDM
  Interventions: Behavioral: Health education on COVID and flu vaccination; Behavioral: Nurse-led shared decision-making; Behavioral: Text messages; Behavioral: Peer navigation
- Experimental Condition 3 (Experimental): Core session, Text messages
  Interventions: Behavioral: Health education on COVID and flu vaccination; Behavioral: Text messages
- Experimental Condition 4 (Experimental): Core session, nurse-led SDM, text messages
  Interventions: Behavioral: Health education on COVID and flu vaccination; Behavioral: Nurse-led shared decision-making; Behavioral: Text messages
- Experimental Condition 5 (Experimental): Core, lottery prize
  Interventions: Behavioral: Health education on COVID and flu vaccination; Behavioral: Lottery prize for vaccination
- Experimental Condition 6 (Experimental): Core session, nurse-led SDM, lottery prize
  Interventions: Behavioral: Health education on COVID and flu vaccination; Behavioral: Nurse-led shared decision-making; Behavioral: Lottery prize for vaccination
- Experimental Condition 7 (Experimental): Core, text messages, lottery prize
  Interventions: Behavioral: Health education on COVID and flu vaccination; Behavioral: Text messages; Behavioral: Lottery prize for vaccination
- Experimental Condition 8 (Experimental): Core, nurse-led SDM, text messages, lottery prize
  Interventions: Behavioral: Health education on COVID and flu vaccination; Behavioral: Nurse-led shared decision-making; Behavioral: Text messages; Behavioral: Lottery prize for vaccination
- Experimental Condition 9 (Experimental): Core, peer navigation
  Interventions: Behavioral: Health education on COVID and flu vaccination; Behavioral: Peer navigation
- Experimental Condition 10 (Experimental): Core, nurse-led SDM, peer navigation
  Interventions: Behavioral: Health education on COVID and flu vaccination; Behavioral: Nurse-led shared decision-making; Behavioral: Peer navigation
- Experimental Condition 11 (Experimental): core, text messages, peer navigation
  Interventions: Behavioral: Health education on COVID and flu vaccination; Behavioral: Text messages; Behavioral: Peer navigation
- Experimental Condition 13 (Experimental): core, lottery prize, peer navigation
  Interventions: Behavioral: Health education on COVID and flu vaccination; Behavioral: Lottery prize for vaccination; Behavioral: Peer navigation
- Experimental Condition 14 (Experimental): core, SDM, lottery prize, peer navigation
  Interventions: Behavioral: Health education on COVID and flu vaccination; Behavioral: Nurse-led shared decision-making; Behavioral: Lottery prize for vaccination; Behavioral: Peer navigation
- Experimental Condition 15 (Experimental): core, text messages, lottery, peer navigation
  Interventions: Behavioral: Health education on COVID and flu vaccination; Behavioral: Text messages; Behavioral: Lottery prize for vaccination; Behavioral: Peer navigation
- Experimental Condition 16 (Experimental): core, SDM, text message, lottery, peer navigation
  Interventions: Behavioral: Health education on COVID and flu vaccination; Behavioral: Nurse-led shared decision-making; Behavioral: Text messages; Behavioral: Lottery prize for vaccination; Behavioral: Peer navigation
- Experimental Condition 2 (Experimental): Core, SDM
  Interventions: Behavioral: Health education on COVID and flu vaccination; Behavioral: Nurse-led shared decision-making

INTERVENTIONS:
Behavioral: Health education on COVID and flu vaccination — 1 session (30 min) with a health educator on vaccination
Behavioral: Nurse-led shared decision-making — 1 session and FU calls with a trained nurse
  Arms: Experimental Condition 10; Experimental Condition 12; Experimental Condition 14; Experimental Condition 16; Experimental Condition 2; Experimental Condition 4; Experimental Condition 6; Experimental Condition 8
Behavioral: Text messages — Health & wellness interactive text message (TM) intervention (12 weeks, 2 texts/week)
  Arms: Experimental Condition 11; Experimental Condition 12; Experimental Condition 15; Experimental Condition 16; Experimental Condition 3; Experimental Condition 4; Experimental Condition 7; Experimental Condition 8
Behavioral: Lottery prize for vaccination — Modest lottery prize for COVID vaccination
  Arms: Experimental Condition 13; Experimental Condition 14; Experimental Condition 15; Experimental Condition 16; Experimental Condition 5; Experimental Condition 6; Experimental Condition 7; Experimental Condition 8
Behavioral: Peer navigation — Peer navigation (4 months duration, contact as needed).
  Arms: Experimental Condition 10; Experimental Condition 11; Experimental Condition 12; Experimental Condition 13; Experimental Condition 14; Experimental Condition 15; Experimental Condition 16; Experimental Condition 9

SUMMARY:
The proposed study responds to the need for community-engaged interventions to increase vaccine uptake among populations experiencing health disparities. We focus on COVID-19 and influenza vaccination, both of which now require annual vaccines. Among those at highest risk for morbidity, hospitalization, and mortality are African American/Black and Latino (ABBL) persons who are not up-to-date on these vaccinations. Only 20-28% of adult AABL persons are up-to-date on COVID-19 vaccination, compared to 31% of White persons, and only 30-40% of AABL persons receive the influenza vaccine annually compared to >55% among White persons. AABL experience serious impediments to COVID-19 (and to a lesser extent, influenza) vaccination at individual- (e.g., distrust, insufficient knowledge, low perceived risk, cognitive biases), social- (e.g., peer norms), and structural-levels of influence (e.g., poor access). Taken together, these comprise multi-level vaccine hesitancy. Factors that promote vaccination include trusted AABL health educators (peers, nurses), tapping into altruism and collective responsibility, circumventing cognitive biases, and reducing structural barriers. Without efforts to address multi-level vaccine hesitancy, rates of COVID-19 and influenza vaccination will remain unacceptably low and racial/ethnic health disparities in infectious disease morbidity and mortality will persist. The proposed study is led by a collaborative team at New York University and the Northern Manhattan Improvement Corporation. It uses the multiphase optimization strategy (MOST), an engineering-inspired framework, to test effects of individual candidate intervention components in a factorial design and then optimize a multi-component intervention made up of the most cost-effective combination of components. Staying up-to-date with COVID-19 vaccination (confirmed with documentary evidence) is the primary outcome, and influenza vaccination is the secondary outcome. We have identified four promising candidate components, with an emphasis on brevity, low-touch, and future scalability: A) nurse-led shared decision making, B) a text message intervention, C) modest lottery prizes for vaccination, and D) peer navigation to vaccination appointments. Participants will be N=560 community-residing adult English and Spanish-speaking AABL persons who are not up-to-date on COVID-19 and influenza vaccinations but with at least one COVID-19 vaccine dose.

DETAILED DESCRIPTION:
The proposed study responds to the need for community-engaged interventions to increase vaccine uptake among populations experiencing health disparities. We focus on COVID-19 and influenza vaccination, both of which now require annual vaccines. Among those at highest risk for morbidity, hospitalization, and mortality are African American/Black and Latino (ABBL) persons who are not up-to-date on these vaccinations. Only 20-28% of adult AABL persons are up-to-date on COVID-19 vaccination, compared to 31% of White persons, and only 30-40% of AABL persons receive the influenza vaccine annually compared to >55% among White persons. AABL experience serious impediments to COVID-19 (and to a lesser extent, influenza) vaccination at individual- (e.g., distrust, insufficient knowledge, low perceived risk, cognitive biases), social- (e.g., peer norms), and structural-levels of influence (e.g., poor access). Taken together, these comprise multi-level vaccine hesitancy. Factors that promote vaccination include trusted AABL health educators (peers, nurses), tapping into altruism and collective responsibility, circumventing cognitive biases, and reducing structural barriers. Without efforts to address multi-level vaccine hesitancy, rates of COVID-19 and influenza vaccination will remain unacceptably low and racial/ethnic health disparities in infectious disease morbidity and mortality will persist. The proposed study is led by a collaborative team at New York University and the Northern Manhattan Improvement Corporation. It uses the multiphase optimization strategy (MOST), an engineering-inspired framework, to test effects of individual candidate intervention components in a factorial design and then optimize a multi-component intervention made up of the most cost-effective combination of components. Staying up-to-date with COVID-19 vaccination (confirmed with documentary evidence) is the primary outcome, and influenza vaccination is the secondary outcome. We have identified four promising candidate components, with an emphasis on brevity, low-touch, and future scalability: A) nurse-led shared decision making, B) a text message intervention, C) modest lottery prizes for vaccination, and D) peer navigation to vaccination appointments. Participants will be N=560 community-residing adult English and Spanish-speaking AABL persons who are not up-to-date on COVID-19 and influenza vaccinations but with at least one COVID-19 vaccine dose. Specific aims are: Aim 1) identify which of four components contribute meaningfully to improvement in the outcomes; Aim 2) identify mediators (e.g., altruism, norms) and moderators (e.g., sociodemographic characteristics, distrust) of the effects of each component; and Aim 3) build the most cost-effective intervention package(s). Participants will be randomly assigned to an experimental condition, and assessed at 3- and 6-months post-baseline; N=45 participants will engage in qualitative in-depth interviews. We will also uncover, describe, and plan for implementation issues so the optimized intervention can be rapidly scaled up by community-based and outpatient health organizations.

ELIGIBILITY:
Inclusion Criteria: 2) can engage in study activities in English or Spanish; 3) Black or African American or Latino/Hispanic race/ethnicity; 4) resides in New York City; 5) has received at least one dose of a COVID-19 vaccination in their lifetime but is not up-to-date on COVID-19 vaccination, defined as has not received the most recently available vaccine, confirmed with documentary evidence; 6) eligible to receive the COVID-19 vaccine (has not had anaphylaxis, myocarditis, pericarditis, or thrombosis with thrombocytopenia syndrome or other adverse effects deemed by a physician to be related to the COVID-19 vaccine) and if previously diagnosed with COVID-19, a minimum of 10 days has elapsed since last test positivity; 7) is not up-to-date on influenza vaccination defined as not yet receiving the available influenza vaccine; 8) has a phone that can be used for study participation and can receive text messages.

-

Exclusion Criteria: NONE

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Vaccination for COVID-19 | 3- and 6-months post-baseline
  Vaccination for COVID-19 with documentary evidence

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-29): https://cdn.clinicaltrials.gov/large-docs/61/NCT06614361/Prot_SAP_000.pdf
  • Informed Consent Form (2025-02-25): https://cdn.clinicaltrials.gov/large-docs/61/NCT06614361/ICF_001.pdf